CLINICAL TRIAL: NCT04058080
Title: Randomized Controlled Trial of Bikram Yoga and Aerobic Exercise for the Treatment of Major Depression: Efficacy and Underlying Mechanisms
Brief Title: Bikram Yoga and Aerobic Exercise for the Treatment of Major Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Queen's University Senate Advisory Research Committee (Unknown)
Responsible Party: Principal Investigator, Dr. Kate Harkness, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSYC-132-13
Record Dates: First submitted 2019-08-01; First posted 2019-08-15 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Depression
Keywords: Major depression; yoga; Bikram yoga; aerobic exercise; complementary and alternative treatment approaches; nontraditional treatment approaches; mindfulness; rumination; stress reactivity; cardiovascular functioning
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Rumination Syndrome | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bikram Yoga (Experimental): Participants in the Bikram yoga group were asked to attend two classes per week for 8 weeks (16 classes in total) at a local affiliated Bikram yoga studio. Certified Bikram yoga teachers instructed all classes using a scripted instructional dialogue. Each 90-min class was held in a temperature-controlled room (40.6 degrees Celsius, 40% humidity). The class opened with a deep breathing exercise and continued with 50 minutes of standing asanas and 40 minutes of floor-based asanas, including a quick, forceful breathing exercise to finish. All but the last asana (i.e., spine-twisting) were performed twice. Savasana, which is a restorative and relaxation posture, was performed between asanas throughout the floor series and at the end of class. The yoga studio regularly offered 22 class times per week, all of which were accessible to participants.
  Interventions: Other: Bikram Yoga
- Aerobic Exercise (Active Comparator): Participants in the aerobic exercise group were asked to attend two group aerobic exercise classes per week for 8 weeks (16 classes in total) at the Kingston Family YMCA. They were provided with a modified schedule of the YMCA group classes, which included only classes with a strong aerobic component and excluded those involving yoga, pilates, or cycling. Selecting these classes was done in consultation with the general manager of the YMCA, who was familiar with each class type. Classes involving the following components were available to participants: choreography-based cardio, aerobics, light muscular conditioning, and stretching; cardio, plyometric, and strength training exercises; high intensity aerobic exercise with intermittent rest periods; circuit-based cardio and strength training exercises; stepper-based exercises; and Latin-inspired dance/fitness. Classes were 50-60 minutes in duration.
  Interventions: Other: Aerobic Exercise
- Waitlist (No Intervention): Waitlisted individuals were not able to access yoga or exercise classes throughout the intervention period but participated in the rest of the study protocol. Following the post-treatment assessment, they received access to the class type of their choosing.

INTERVENTIONS:
Other: Bikram Yoga — Participants in the Bikram yoga group were asked to attend two classes per week for 8 weeks (16 classes in total) at a local affiliated Bikram yoga studio. Certified Bikram yoga teachers instructed all classes using a scripted instructional dialogue. Each 90-min class was held in a temperature-controlled room (40.6C, 40% humidity). The yoga studio regularly offered 22 class times per week, all of which were accessible to participants.
  Arms: Bikram Yoga
Other: Aerobic Exercise — Participants in the aerobic exercise group were asked to attend two group aerobic exercise classes per week for 8 weeks (16 classes in total) at the Kingston Family YMCA. They were provided with a modified schedule of the YMCA group classes, which included only classes with a strong aerobic component and excluded those involving yoga, pilates, or cycling. Classes involving the following components were available to participants: choreography-based cardio, aerobics, light muscular conditioning, and stretching; cardio, plyometric, and strength training exercises; high intensity aerobic exercise with intermittent rest periods; circuit-based cardio and strength training exercises; stepper-based exercises; and Latin-inspired dance/fitness. Classes were 50-60 minutes in duration. Participants were able to attend any of the offered classes each week. Participants had approximately 18-22 classes in total to choose from each week.
  Arms: Aerobic Exercise

SUMMARY:
The primary goal of this project was to examine the antidepressant effects of yoga as an alternative treatment for depression as compared to no treatment and aerobic exercise. The secondary goal of this project was to examine relevant physiological (i.e., heart rate, blood pressure, cortisol levels) and psychological variables (i.e., perceived hassles, rumination, mindfulness) that may underlie the antidepressant effects of Bikram yoga and aerobic exercise.

DETAILED DESCRIPTION:
Participants attended two pre-treatment appointments. The first pre-treatment appointment was a 2-hour psychological assessment in which the study and its protocol were explained at length and consent was collected. Participants then completed a battery of measures, including a medical screening interview, a demographic interview, the full Structured Clinical Interview for DSM-IV Axis I Disorders, and the Hamilton Rating Scale for Depression. Participants also completed self-report psychological measures during the psychological assessment. After completion of this appointment, participants were given instructions to avoid specific substances or activities for a minimum length of time before the second pre-treatment appointment.

The second pre-treatment appointment was a 3-hour physiological assessment which was completed within 1 week of the psychological assessment. The first 30 minutes of this appointment were used to set-up the physiological measurements and allow enough time for participants to become familiarized and comfortable with the laboratory setting. Following this, a carefully timed experimental protocol was followed, during which heart rate and mean arterial pressure were measured and recorded continuously. The participants also completed a stress task and their saliva was collected. The participants also engaged in the Submaximal Cycle Ergometer Test. At the end of the physiological assessment, participants were randomly assigned via a computer-generated random sequence to one of the treatment conditions. Group assignment was revealed via sealed envelopes that had been previously prepared by research personnel. Participants who were in the waitlist group were offered yoga or aerobic classes after the completion of the study protocol.

Participants in the yoga and aerobic exercise groups then attended 2 classes per week of either yoga or aerobic exercise for 8 weeks.

Following completion of the intervention period, participants attended a 3½ hr post-treatment assessment in which all measures of the physiological pre-treatment assessment were repeated. Additionally, participants were administered the Mood Module of the SCID-I/P and the HAM-D to assess changes in diagnostic status and depression severity.

ELIGIBILITY:
Inclusion Criteria:

* Physically healthy
* Female
* Meet DSM-IV-TR criteria for a current episode of a non chronic, unipolar depressive disorder (i.e., MDD, adjustment disorder with depressed mood, depressive disorder not otherwise specified)

Exclusion Criteria:

* Presence of a psychotic disorder, bipolar disorder, substance dependence, current suicidality beyond simple ideation
* Presence of a medical condition that could be the cause of depression
* Presence of a a pre-existing physical condition that could interfere with participation in physical activity (e.g., cardiovascular disease, untreated hypertension, etc.)
* Change in the type or dose of antidepressant medication or change in frequency of sessions of psychotherapy/counseling in the previous 3 months
* Pregnant women or women actively trying to become pregnant
* Regular participation in yoga or group exercise classes (i.e., on a biweekly or more basis) during the 3-month period prior to study onset or on a long-term basis in the past 2 years
* A schedule that did not allow for participation in yoga or exercise classes twice per week

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2013-03-12 (Actual); Primary Completion 2016-03-13 (Actual); Study Completion 2016-03-13 (Actual)

PRIMARY OUTCOMES:
Treatment Response | Psychological pre-treatment assessment, post-treatment assessment (upon completion of 8 week intervention)
  Treatment response was defined as a 50% reduction from pre-treatment assessment and post-treatment assessment on the Hamilton Rating Scale for Depression (HAM-D). The HAM-D is a 17-item semi-structured interview that assesses the severity of depressive symptoms in the past week. The item ratings range from 0 to 2 or from 0 to 4 depending on the item, with total scores ranging from 0 to 50. Higher scores indicate more severe depressive symptoms.
Depression remission | Post-treatment assessment (upon completion of 8 week intervention)
  Remission was defined according to two criteria:
  1. A post-treatment assessment Hamilton Rating Scale for Depression (HAM-D) score of 7 or lower. The HAM-D is a 17-item semi-structured interview that assesses the severity of depressive symptoms in the past week. The item ratings range from 0 to 2 or from 0 to 4 depending on the item, with total scores ranging from 0 to 50. Higher scores indicate more severe depressive symptoms.
     AND
  2. No longer meeting diagnostic criteria for major depression. This was assessed by administering the major depression module of the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-I/P). The major depression module of the SCID-I/P includes 9 questions corresponding to the 9 criterial symptoms of major depression. Each symptom is coded as 0-absent or 1-present. Total scores can range from 0-9. A total score of 5 or above indicates the presence of major depression. Scores below 5 indicate that the participant no longer meets criteria.

SECONDARY OUTCOMES:
Hassles and Uplifts Scale (HUS) | Psychological pre-treatment assessment, throughout intervention period (weekly for the 8 weeks of intervention)
  The Hassles and Uplifts Scale (HUS) examines commonly encountered events that may be considered irritants (i.e., hassles) and/or positive experiences (i.e., uplifts). More specifically, participants were asked to give weekly ratings of 53 events based on how much each event was a hassle and how much each event was an uplift in the previous week with the following scale: 0 = None or not applicable, 1 = Somewhat, 2 = Quite a bit, 3 = A great deal. Scores across items were summed to give separate cumulative scores for hassles and uplifts. For the purposes of this study, only hassles were examined in subsequent analyses. The range of possible scores for hassles is 0 to 159, with a higher score indicating greater hassles.
Ruminative Responses Scale (RRS) of the Response Styles Questionnaire | Psychological pre-treatment assessment, throughout intervention period (bi-weekly for the 8 weeks of intervention)
  The Ruminative Responses Scale (RRS) of the Response Styles Questionnaire was administered to assess the tendency to ruminate in response to depressive symptoms. The RRS has 22 items, rated on a 4-point scale ranging from 1 (almost never) to 4 (almost always) and asks respondents to indicate what they "generally do when feeling down, sad, or depressed". In this study, instructions were modified slightly in that participants were asked to indicate their general tendencies within a specific time frame (i.e., during the past 2 weeks). An overall score was computed by summing responses across all items. The range of possible scores on this scale is 22 to 88, with a higher score indicating more rumination.
Philadelphia Mindfulness Scale (PHLMS) | Psychological pre-treatment assessment, throughout intervention period (weekly for 8 weeks of intervention classes)
  The 20-item Philadelphia Mindfulness Scale (PHLMS) was used to asses two components of mindfulness, present-moment awareness and acceptance. Participants responded to each item on 5-point scale, ranging from 1 (Never) to 5 (Very Often). Scores across items were summed to give separate cumulative scores for awareness and acceptance. Prior to calculating the acceptance score, all acceptance-related items were reverse coded. Scores for awareness and acceptance range from 10 to 50, with higher scores indicate higher awareness or acceptance.
Heart Rate | Physiological pre-treatment assessment (within 30 minutes of start), post-treatment assessment (upon completion of 8 week intervention)
  Heart rate (HR) was assessed using three ECG electrodes on the chest and abdomen.
Blood Pressure | Physiological pre-treatment assessment (within 30 minutes of start), post-treatment assessment (upon completion of 8 week intervention)
  Mean arterial pressure (MAP) was assessed using an automated blood pressure device called a finger photoplethysmography.
Stress Sensitivity: Salivary Hormone and Trier Social Stress Test (TSST) | Physiological pre-treatment assessment (~30 minutes into the protocol), post-treatment assessment (upon completion of 8 week intervention)
  Participants were required to explain why they deserved a particular job opportunity after being recently fired or defend themselves against a false accusation of shoplifting. Immediately following the speech task, participants underwent a mental arithmetic task in which they were asked to serially subtract 13 from a 4-digit prime number. Saliva samples were collected 8 times throughout the test.
Submaximal Exercise Test | Physiological pre-treatment assessment (after TSST), post-treatment assessment (upon completion of 8 week intervention)
  In this test, participants exercised on a cycle ergometer while their heart rate was monitored. This test was used to estimate maximal oxygen uptake.

CONTACTS AND LOCATIONS:
Overall Officials: Kate Harkness, PhD, Principal Investigator — Queen's University

IPD SHARING:
Plan to Share IPD: No